CLINICAL TRIAL: NCT00643461
Title: Clinical Evaluation of Three Dental Adhesive Systems in Class V Restorations
Status: Completed | Type: Observational
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Other Study IDs: CR-07-009
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Adhesive A
  Interventions: Device: Adhesive A
- Adhesive B
  Interventions: Device: Adhesive B
- Adhesive C
  Interventions: Device: Adhesive C

INTERVENTIONS:
Device: Adhesive A — Applied per manufacturer's instructions.
  Other Names: Adper Scotchbond SE (3M ESPE)
  Groups: Adhesive A
Device: Adhesive B — Applied per manufacturer's instructions.
  Other Names: Adper Easy Bond (3M ESPE)
  Groups: Adhesive B
Device: Adhesive C — Applied per manufacturer's instructions.
  Other Names: Single Bond Plus (3M ESPE)
  Groups: Adhesive C

SUMMARY:
The purpose of this study is to compare the clinical performance of three dental adhesive systems used to bond Class V cavity fillings in adult teeth.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 19 years of age
* Must have at least 3 qualifying noncarious Class V lesions of appropriate depth
* Must be willing to sign consent form
* Must be willing and able to return to UAB clinic for 4 study appointments
* Must be in good medical health and able to tolerate dental procedures

Exclusion Criteria:

* Current participation in other restorative product studies
* Severe salivary gland dysfunction
* Rampant caries (cavities)
* Chronic periodontitis (gum disease)
* Known allergies to the study materials
* Unacceptable level of oral hygiene
* Inability or unwillingness to attend study appointments

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Class V cavities
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2008-04; Primary Completion 2012-02 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Retention of the restoration. | 6, 12, 24, 36 months post-placement

CONTACTS AND LOCATIONS:
Overall Officials: John O Burgess, MS, DDS, Principal Investigator — University of Alabama at Birmingham (UAB) School of Dentistry
Locations (1):
- University of Alabama at Birmingham (UAB) School of Dentistry, Birmingham, Alabama, United States